CLINICAL TRIAL: NCT06563193
Title: Urinary Neurotrophin Levels as Potential Biomarkers for Overactive Bladder: A Case-Control Study
Acronym: urinary
Status: Enrolling by invitation | Type: Observational
Sponsor: Erzincan Binali Yildirim Universitesi (Other)
Responsible Party: Principal Investigator, OZGUR EKICI, Assistant Professor, Erzincan Binali Yildirim Universitesi
Other Study IDs: ERZ-OE-01
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- overactive bladder group: OAB was diagnosed according to the patient's complaint of urgency with or without urge incontinence as the core symptom according to the criteria defined by the International Continence Society
- control group: As a control group, patients who were admitted to the outpatient clinic for other reasons and who did not have OAB symptoms and have normal voiding functions were included
  Interventions: Diagnostic Test: NERVE GROWTH FACTOR

INTERVENTIONS:
Diagnostic Test: NERVE GROWTH FACTOR — urinary neurotrophins
  Other Names: BRAIN DERIVED NEUROTRPHIC FACTOR
  Groups: control group

SUMMARY:
Overactive bladder is a prevalent urological disorder marked by symptoms such as urinary urgency, increased frequency of urination, and nighttime urination (nocturia). Neurotrophins, including nerve growth factor and brain-derived neurotrophic factor, play crucial roles in the development and function of neurons. Recent research has suggested a possible connection between these neurotrophins and OAB.

This study sought to explore the relationship between urinary levels of NGF and BDNF and the presence of OAB.

DETAILED DESCRIPTION:
Ethics committee approval dated 22.02.2024 and numbered 2024-03/01 was obtained from Erzincan Binali Yıldırım University Faculty of Medicine Ethics committee for the study.

Between February 2024 and July 2024, patients between the ages of 18 and 75 who were admitted to the urology outpatient clinic with a preliminary diagnosis of OAB and diagnosed with OAB were prospectively included in the study. Patients were asked to complete a 3-day voiding diary. OAB was diagnosed according to the patient's complaint of urgency with or without urge incontinence as the core symptom according to the criteria defined by the International Continence Society. The study was conducted in accordance with the principles of the 2008 Helsinki Declaration.

Demographic data including age, gender and BMI were recorded. With the OAB-V8 questionnaire scores (0-40), Indevus Urgency Severity Scale (IUSS) scores, the number of urgency, pollakiuria and nocturia episodes were also recorded. The OAB-V8 questionnaire is a form consisting of 8 questions with each question being scored between 0-5 and a total score of 40 points. A total score above 8 is considered significant [7]. Indevus Urgency Severity Scale (IUSS) classified as 0-4, representing no urgency, occasional urgency which was always tolerable, urgency which was tolerable for 5 min, urgency which was intolerable, and urgency which was usually accompanied by incontinence, respectively [6, 8]. Blood group, creatitine values from peripheral blood and urine samples were recorded at outpatient clinic visits. BDNF and NGF levels were measured from the urine samples taken at the patients' outpatient clinic admissions. Urine samples were studied before treatment was given. Informed consent was obtained from all participants before urine was collected.

Patients with urinary tract infection, systemic inflammation, renal function test disorders, patients with a history of previous urological surgery, patients with a history of urological malignancy, patients with bladder stones, benign prostatic hyperplasia and urethral stricture were excluded from the study. As a control group, patients who were admitted to the outpatient clinic for other reasons and who did not have OAB symptoms and have normal voiding functions were included. Urine samples of these patients were also recorded.

Urine samples were collected from both OAB subjects and controls. Urine was collected in sterile specimen jars, transferred to sterile test tubes, and frozen at 80.8C. The samples were then thawed and centrifuged at 200 relative centrifugal force for 5 min. The supernatant was aliquoted and stored at 80.8C until further processing. A 3-ml urine sample was obtained concurrently for measuring urinary creatinine (Cr) levels. Urine samples were used for Human Brain Derived Neurotrophic Factor (BDNF) and Human Nerve Growth Factor (NGF) levels. The kits were used to test the level of BDNF (Shanghai Coon Koon Biotech Co., Ltd China. Cat No:CK-bio-10643) and NGF (Shanghai Coon Koon Biotech Co., Ltd China. Cat No:CK-bio-12600) based on the principle of double antibody sandwich technology enzyme linked immunosorbent assay (ELISA). The analytical (linear) detection range for BDNF was 1-24 ng/mL. The minimal detection limit for BDNF was 0.1 ng/mL . The analytical (linear) detection range for NGF was 10-160 pg/mL. The minimal detection limit for NGF was 1.0 pg/mL.

The data recorded at baseline were compared between the groups.

ELIGIBILITY:
Inclusion Criteria: adult patients (aged 18-75 years) presenting to the urology outpatient clinic with a preliminary OAB diagnosis -

Exclusion Criteria:

-

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult patients (aged 18-75 years) presenting to the urology outpatient clinic with a preliminary OAB diagnosis
  -
Sampling Method: Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
NGF anf BDNF levels in overactive bladder patients | 6 months
  NGF AND BDNF LEVELS ARE HIGH IN PATIENTS WITH OVERACTIVE BLADDER.

CONTACTS AND LOCATIONS:
Overall Officials: Ozgur EKICI, Study Chair — ErzincanBinaliYildirim
Locations (1):
- Erzincan Binali Yıldırım University, Erzincan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No